CLINICAL TRIAL: NCT07258901
Title: Optimizing Postoperative Pain Management After Percutaneous Nephrolithotomy: A Comparative Clinical Assessment
Brief Title: Postoperative Analgesia Practices After Percutaneous Nephrolithotomy
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, assoc prof, Istinye University
Other Study IDs: 231-2025
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Nephrolithiasis
Keywords: Percutaneous Nephrolithotomy; Postoperative Analgesia; Pain Management; Regional Anesthesia; Nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- quadro iliac plane block: quadro iliac plane block
- erector spinae nerve block: erector spinae nerve block
- Intravenous opioid-based analgesia: Intravenous opioid-based analgesia

SUMMARY:
This prospective observational study aims to evaluate the effectiveness and safety of different postoperative analgesia methods used in patients undergoing percutaneous nephrolithotomy (PCNL). Analgesia techniques are determined independently by the responsible anesthesiologist as part of routine clinical practice, and the study team does not intervene in treatment decisions.

DETAILED DESCRIPTION:
This is a prospective observational clinical study designed to examine the impact of various postoperative analgesia strategies on pain outcomes in patients undergoing percutaneous nephrolithotomy (PCNL). In routine practice at the participating center, regional block techniques and intravenous analgesia protocols are commonly used, and different anesthesiologists may choose different postoperative analgesia approaches.

All patients will undergo standard general anesthesia according to institutional protocols. Intraoperative monitoring will include heart rate, mean arterial pressure, oxygen saturation, duration of surgery, opioid consumption, and intraoperative complications. Postoperative follow-up will include assessment of pain scores (NRS) at 0, 2, 6, 12, and 24 hours, cumulative opioid consumption, need for rescue analgesics, time to first analgesic request, incidence of postoperative nausea and vomiting (PONV), antiemetic use, patient satisfaction, and any analgesia-related adverse events.

Demographic characteristics (age, sex, BMI, ASA status), stone features (location, side, volume), and intraoperative variables will be recorded. Data will be collected prospectively and stored securely.

The primary goal is to compare the effect of different postoperative analgesia methods on cumulative opioid use in the first 24 hours. Secondary aims include evaluating pain scores, rescue analgesic need, intraoperative opioid use, time to first analgesic request, PONV incidence, patient satisfaction, and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* ASA physical status I-III
* Undergoing unilateral PCNL
* Providing written informed consent

Exclusion Criteria:

* Known allergy to local anesthetics

Coagulopathy or contraindication to regional anesthesia

BMI > 35 kg/m²

Cognitive or communication impairment affecting pain evaluation

Neurological or psychiatric disorders

Musculoskeletal abnormalities

Chronic opioid use, alcohol or substance abuse history

Previous PCNL or open renal surgery on the same side

Refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 65 years undergoing unilateral percutaneous nephrolithotomy (PCNL) at Haseki Training and Research Hospital. All participants are ASA physical status I-III and receive postoperative analgesia according to routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-02 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption | 24 hours
  Cumulative opioid consumption in the first 24 hours

SECONDARY OUTCOMES:
Pain scores at rest and during movement | 0, 2, 6, 12, and 24 hours postoperatively
  Pain intensity measured using the Numeric Rating Scale (NRS), a validated 11-point pain scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Higher scores represent worse pain
Time to first analgesic request | Postoperative 24 hours
  Time to first analgesic request
Need for rescue analgesics | 24 hours
  Need for rescue analgesics
Intraoperative opioid consumption | During surgery
  Intraoperative opioid consumption
Antiemetic medication use | 24 hours
  Antiemetic medication use
Patient satisfaction score | 24 hours postoperatively
  Patient satisfaction regarding postoperative analgesia, assessed using a Numeric Rating Scale (NRS) ranging from 0 to 10, where 0 represents no satisfaction and 10 represents the highest possible satisfaction. Higher scores indicate better satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.